CLINICAL TRIAL: NCT01065610
Title: Oxytocin Buffers Cortisol Responses to Stress in Individuals With Impaired Coping Abilities
Brief Title: Oxytocin Buffers Stress Response in Individuals With Impaired Coping Abilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Osnabrueck (Other)
Other Study IDs: Neurolab_RD_001
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Last update posted 2010-02-09 (Estimated); Status verified 2010-01

CONDITIONS: Coping Skills; Oxytocin; Stress
MeSH Terms: interventions — Oxytocin

ARMS (2):
- Oxytocin (Experimental): Intranasal Oxytocin, 24 IU
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin
  Arms: Oxytocin
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study investigated, if people with impaired coping abilities benefit from intranasal oxytocin application.

ELIGIBILITY:
Inclusion Criteria:

* male

Exclusion Criteria:

* psychological disorders
* drug abuse
* cigarette smoking
* coronary diseases
* nervous system diseases

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2008-01; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Salivary Cortisol